CLINICAL TRIAL: NCT06825455
Title: Clinical Study of the Safety and Tolerability of B7H3 CAR-γδT Cell Injection in the Treatment of Advanced Solid Tumors
Brief Title: Allogeneic B7H3 CAR-γδT Cell Therapy for Advanced Solid Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Vice President of Beijing Cancer Hospital, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH10407-ST-01（0）
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors; Ovarian Cancers; Peritoneal (metastatic) Cancer
Keywords: cell therapy; γδT; CAR-T
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Masking Description: Patients with B7H3-positive advanced solid tumors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous infusion groups (Experimental): Patients with advanced solid tumor. A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, allogenic targeting B7H3 chimeric antigen receptor γδT cells.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: B7H3 CAR-γδT cells
- Abdominal infusion group (Experimental): Patients with ovarian cancer or peritoneal (metastatic) cancer.Before cell injection, for subjects with obvious ascites, the ascites should be pumped as clean as possible through peritoneal puncture, and then the abdomen should be rinsed with saline before the cell infusion is performed.
  Interventions: Biological: B7H3 CAR-γδT cells

INTERVENTIONS:
Drug: Fludarabine — Intravenous infusion group:30mg/m2 x 3 days (Day-4~-2)
  Arms: Intravenous infusion groups
Drug: Cyclophosphamide — Intravenous infusion group:500mg/m2 x 3 days (Day-4~-2)
  Arms: Intravenous infusion groups
Biological: B7H3 CAR-γδT cells — A single infusion of 6.0×107 CAR+ cells, 2.0×108CAR+ cells, and 6.0×108CAR+ cells

SUMMARY:
γδT cells can directly recognize non-peptide tumor antigens, such as IPP phosphorylated metabolites, without relying on specific major histocompatibility complexes (MHCs). This unique characteristic leads to a lower risk of graft-versus-host disease (GVHD). The clinical safety of γδT cells in allogeneic tumor therapies has been validated multiple times, highlighting their significant potential in developing universal CAR-T cell therapies.

B7H3 (CD276), a member of the B7 negative co-stimulatory molecule family, is minimally expressed or absent in normal tissues but highly expressed in various tumor tissues. As a result, B7H3 is regarded as a highly promising tumor-associated antigen and a universal drug target with substantial therapeutic potential.

By utilizing γδT cells as carrier cells, the development of universal B7H3 CAR-γδT cell injections for advanced solid tumors can effectively address risks such as autologous cell preparation failure and treatment delays. This innovative approach offers a highly efficient solution for solid tumor treatment and holds great promise for advancing immunotherapy in this field

DETAILED DESCRIPTION:
This study is an open-label, dose-escalation exploratory clinical trial using γδ T cells derived from healthy donors, genetically engineered to express a chimeric antigen receptor (CAR) targeting B7H3 on their membrane. Preclinical in vitro and in vivo experiments demonstrated the modified CAR-γδ T cells possess specific cytotoxicity against B7H3-positive tumor cells.

According to the patients' disease conditions, they were divided into an intravenous infusion group and an intraperitoneal infusion group. Both groups underwent a dose-escalation study using the "3+3" design.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited;
2. Expected survival time ≥3 months;
3. ECOG score 0~1;
4. Patients who meet the clinical diagnostic criteria and have a clear pathological diagnosis of malignant solid tumors that have failed standard treatment;
5. Tumor tissue samples (specimens within one year are recommended) positive for B7H3 by immunohistochemical (IHC) staining or flow assay;
6. Presence of at least one evaluable lesion according to RECIST V1.1;
7. Tumors limited to peritoneal (metastatic) and ovarian cancer in patients in the laparotomy group;
8. Substantially normal bone marrow reserve function and normal liver and renal function (laboratory tests need to be fulfilled before the first treatment with cell injection):

   Blood: white blood cell count (WBC) ≥3E9/L, lymphocyte count (LY) ≥0.8E9/L, hemoglobin (Hb) ≥80g/L, platelet (PLT) ≥75E9/L; Liver: ALT ≤ 3 × ULN; AST ≤ 3 × ULN; total bilirubin ≤ 3.0 × ULN; Kidney: serum creatinine ≤ 1.5 × upper limit of normal range (ULN); Heart: left ventricular ejection fraction ≥50% on echocardiography; lung: normal oxygen saturation without oxygen.
9. Pregnancy test should be negative for women of childbearing potential and both men and women agree to use effective contraception during treatment and for 1 year thereafter;
10. Be able to understand the requirements and matters of the trial and be willing to participate in the clinical study as required;
11. Sign the trial informed consent form.

Exclusion Criteria:

1. Known hypersensitivity, allergy, intolerance, or contraindication to cell infusion or any of the drug components that may be used in the study, including fludarabine and cyclophosphamide;
2. Patients who have been continuously using immunosuppressive drugs within 1 month prior to cell infusion;
3. Cerebrovascular accident or seizure within 6 months prior to signing the informed consent form;
4. Symptomatic brain metastases;
5. a known psychiatric or substance abuse disorder that would interfere with cooperation with the trial requirements;
6. Hepatitis B surface antigen (HBsAg) positivity or hepatitis B core antibody (HBcAb) positivity and a peripheral blood test for hepatitis B virus (HBV) DNA titer that is not within the normal reference range; hepatitis C virus (HCV) antibody positivity and peripheral blood hepatitis C virus (HCV) RNA positivity; human immunodeficiency virus (HIV) antibody positivity; syphilis Positive for syphilis;
7. Serious cardiac disease: including, but not limited to, unstable angina pectoris, myocardial infarction (occurring within 6 months prior to screening), congestive heart failure (NYHA classification ≥ III), and severe arrhythmias;
8. Presence of active or uncontrolled infections requiring systemic therapy (except for mild genitourinary and upper respiratory tract infections);
9. has not recovered from acute toxic effects of prior therapy (prior therapy-induced hematologic or organ toxicity ≥ Grade 2, except for abnormalities related to study disease and medical history);
10. have a confirmed diagnosis of an immunodeficiency
11. suffering from an active infection requiring systemic therapy;
12. a female subject of childbearing potential who plans to become pregnant within 2 years of cell infusion; or a male subject whose partner plans to become pregnant within 2 years of cell infusion;
13. Participation in a clinical study of another innovative drug within 1 month prior to screening;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of randomization to 12 months after B7H3 CAR-γδT cells infusion. Among them, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria, graft-versushost disease (GVHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Best objective Response Rate | 12 months
  The incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as the best response to treatment assessed by investigators and based on the RECIST 1.1 criterion.
Duration of Response (DOR) | 12 months
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators and based on the RECIST 1.1 criterion, or death regardless of cause.
Progression Free Survival (PFS) | 12 months
  PFS is defined as the time from the B7H3 CAR-γδT cells infusion date to the date of disease progression assessed by investigators and based on the RECIST 1.1 criterion, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Overall Survival (OS) | 12 months
  OS is defined as the time from B7H3 CAR-γδT cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Immunogenicity: Proportion of subjects with anti drug antibody (ADA) | 12 months
  ADAs include anti-donor γδT antibody or anti-B7H3 CAR single-chain variable fragment antibody.
Pharmacodynamics | Up to 28 days after infusion
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP), ferritin. Peak was defined as the maximum post-baseline level of the cytokine.
Pharmacokinetics | 12 months
  Persistence of B7H3 CAR-γδT cell assessed by number in peripheral blood and ascites

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No